CLINICAL TRIAL: NCT00989729
Title: Preoperative Methylprednisolone in Endovascular Aortic Repair - a Randomized Double Blind Placebo Controlled Clinical Trial
Brief Title: Preoperative Methylprednisolone in Endovascular Aortic Repair
Acronym: POMEVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louise de la Motte (Other)
Responsible Party: Sponsor-Investigator, Louise de la Motte, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVAR-150-2009; EudraCT number 2009-013441-28; H-A-2009-043
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Endovascular Aortic Repair; Methylprednisolone; Systemic inflammatory response syndrome
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Systemic Inflammatory Response Syndrome | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): 75 patients will receive a single preoperative dosage of Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Physiological Saline (Placebo Comparator): 75 patients will receive a single preoperative dosage of Physiological Saline
  Interventions: Drug: Physiological Saline

INTERVENTIONS:
Drug: Methylprednisolone — A single preoperative dosage 30 mg/kg Methylprednisolone suspended in physiological saline (100 ml in total) given intravenously as a 30 minute infusion, 2 hours before surgery.
  Other Names: Solu-Medrol, Pfizer.
  Arms: Methylprednisolone
Drug: Physiological Saline — A single preoperative dosage 100 ml given intravenously as a 30 minute infusion, 2 hours before surgery
  Other Names: Physiological Saline 9 mg/ml, Fresenius Kabi
  Arms: Physiological Saline

SUMMARY:
The purpose of this study is to attenuate the systemic inflammatory response after Endovascular repair of abdominal aortic aneurysms, by administration of a single preoperative dosage of Methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Elective endovascular repair of an asymptomatic abdominal aortic aneurysm.
* Informed signed consent

Exclusion Criteria:

* Positive HIV status, positive hepatitis B or C status
* Immunoinflammatory disease - except topically treated skin disease and respiratory disease.
* Glaucoma
* Gastric or duodenal ulcer
* Systemic fungal infection
* Immunosuppressive treatment
* Current treatment for cancer
* Allergy towards contents of Solu-Medrol
* Alcohol consumption: Men > 21 drinks and women > 14 drinks weekly
* Pregnancy
* Lack of informed signed consent
* Patients where follow up is planned at other location than Rigshospitalet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Systemic inflammatory response syndrome - SIRS | Within 5 postoperative days

SECONDARY OUTCOMES:
Length of postoperative hospital stay | Until discharge
Interleukin 6 plasma level | Within 5 postoperative days
Adverse events related to Methylprednisolone | Within 5 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Louise de la Motte, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Vascular Surgery, Rigshospitalet 3111, Copenhagen, Denmark

REFERENCES:
- [Result] de la Motte L, Kehlet H, Vogt K, Nielsen CH, Groenvall JB, Nielsen HB, Andersen A, Schroeder TV, Lonn L. Preoperative methylprednisolone enhances recovery after endovascular aortic repair: a randomized, double-blind, placebo-controlled clinical trial. Ann Surg. 2014 Sep;260(3):540-8; discussion 548-9. doi: 10.1097/SLA.0000000000000895. PMID 25115430